CLINICAL TRIAL: NCT02642991
Title: Dispensing Study for The Phenacite Project
Brief Title: Dispensing Study for a New Study Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-15-41; NCT02642341 (obsolete NCT alias); NCT02642354 (obsolete NCT alias)
Record Dates: First submitted 2015-12-07; First posted 2015-12-30 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Phenacite Test lens then comfilcon A control lens (Experimental): Participants were randomized to wear Phenacite test lens for one week then cross-over to wear comfilcon A control lens for one week.
  Interventions: Device: Phenacite; Device: comfilcon A
- Comfilcon A control lens then Phenacite test Lens (Active Comparator): Participants were randomized to wear comfilcon A control lens for one week then cross over to Phenacite test lens for one week.
  Interventions: Device: Phenacite; Device: comfilcon A

INTERVENTIONS:
Device: Phenacite — contact lens
Device: comfilcon A — contact lens

SUMMARY:
This study investigated the performance criteria over one week of daily wear to determine if the comfilcon A asphere lens (test) performed equivalently to the comfilcon A sphere (control) in terms of measurement and subjective ratings of visual performance.

DETAILED DESCRIPTION:
This study was a prospective, single site, daily wear, double masked, randomized bilateral cross over dispensing study of binocular wear of comfilcon A asphere lens (test) and comfilcon A sphere lens (control) over 1 week of daily wear.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Oculo-visual examination in the last two years
* Between 18 and 35 years of age and has full legal capacity to volunteer
* Has read and understood the informed consent letter
* Is willing and able to follow instructions and maintain the appointment schedule
* Is correctable to a visual acuity of 20/25 or better (in each eye) with their habitual correction or 20/20 best corrected
* Currently wears, or has previously successfully worn, soft contact lenses between -1.00D (Diopoter) and -4.00D
* Spherical Contact Lens Rx between -1.00 and -4.00 and spectacle cylinder <-0.75
* Has not worn lenses for at least 12 hours before the initial visit
* Has a subjective response at baseline, which indicates suitability for this study
* Currently spends a minimum of 4 hours a day; 5 days a week on digital devices and can replicate this time during the study period
* Is willing and able to wear the study contact lenses a minimum of 10 hours per day; 5 days a week

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has never worn contact lenses before
* Any systemic disease affecting ocular health
* Is using any systemic or topical medications that will affect ocular health
* Has known sensitivity to the diagnostic pharmaceuticals or study products used in this study.
* Has any ocular pathology or anomaly that would affect the wearing of the lenses
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye
* Is aphakic
* Has anisometropia of >1.00
* Has undergone corneal refractive surgery
* Has strabismus
* Has any ocular amblyopia >= 1line of HC (High Contrast) Visual Acuity
* Is participating in any other type of eye related clinical or research study
* Has previously participated in study of the Phenacite lenses

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, Principal Investigator — CCLR, University of Waterloo; Pete Kollbaum, OD, PhD, Principal Investigator — CORL, Indiana University; Meng Lin, OD, PhD, Principal Investigator — CRC, University of California, Berkeley
Locations (3):
- United States (2):
  - University of California, Berkeley, California
  - CORL, Indiana University, Bloomington, Indiana
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | Phenacite Test Lens Then Comfilcon A Control Lens | Comfilcon A Control Lens Then Phenacite Test Lens
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Phenacite Test Lens Then Comfilcon A Control Lens | Comfilcon A Control Lens Then Phenacite Test Lens
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear phenacite study lens and comfilcon A control lens for one week.
Arm/Group | Overall Study
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.1 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 16
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (VA) - High Illumination
Description: Distance visual acuity High Illumination was assessed using logMAR
Time Frame: Baseline (after 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Phenacite Test Lens: Participants were randomized to wear Phenacite test lens for one week
  Phenacite: contact lens
- Comfilcon A Control Lens: Participants were randomized to wear comfilcon A control lens for one week
  comfilcon A: contact lens
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
logMAR
  Monocular | -0.10 (0.07) | -0.11 (0.08)
  Binocular | -0.15 (0.06) | -0.17 (0.07)

2. Primary Outcome: Distance Visual Acuity (VA) - High Illumination
Description: Distance visual acuity High Illumination was assessed using logMAR
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
logMAR
  Monocular | -0.10 (0.08) | -0.11 (0.08)
  Binocular | -0.15 (0.07) | -0.16 (0.06)

3. Primary Outcome: Near Visual Acuity (VA) - High Illumination
Description: Near Visual Acuity (VA) - High Illumination assessed using logMAR
Time Frame: Baseline (after 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
logMAR
  Monocular | -0.07 (0.09) | -0.08 (0.08)
  Binocular | -0.13 (0.09) | -0.14 (0.08)

4. Primary Outcome: Near Visual Acuity (VA) - High Illumination
Description: Near Visual Acuity (VA) - High Illumination assessed using logMAR
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
logMAR
  Monocular | -0.06 (0.10) | -0.07 (0.09)
  Binocular | -0.11 (0.09) | -0.13 (0.10)

5. Primary Outcome: Distance Visual Acuity (VA) - Low Illumination
Description: Distance Visual Acuity (VA) - Low Illumination assessed using logMAR
Time Frame: Baseline (after 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
logMAR
  Monocular | 0.07 (0.08) | 0.05 (0.08)
  Binocular | 0.02 (0.06) | 0.00 (0.06)

6. Primary Outcome: Distance Visual Acuity (VA) - Low Illumination
Description: Distance Visual Acuity (VA) - Low Illumination assessed using logMAR
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
logMAR
  Monocular | 0.06 (0.08) | 0.05 (0.10)
  Binocular | -0.01 (0.06) | 0.01 (0.07)

7. Primary Outcome: Near Visual Acuity (VA) - Low Illumination
Description: Near Visual Acuity (VA) - Low illumination assessed using logMAR
Time Frame: Baseline (after 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
logMAR
  Monocular | 0.15 (0.16) | 0.14 (0.15)
  Binocular | 0.10 (0.16) | 0.08 (0.15)

8. Primary Outcome: Near Visual Acuity (VA) - Low Illumination
Description: Near Visual Acuity (VA) - Low illumination assessed using logMAR
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
logMAR
  Monocular | 0.16 (0.17) | 0.18 (0.17)
  Binocular | 0.09 (0.16) | 0.11 (0.17)

9. Primary Outcome: Quality of Distance Vision
Description: Subjective scoring of Quality of Distance Vision assessed using 0-100 continuous scale: (0=extremely poor vision all of the time. 100=excellent vision all of the time)
Time Frame: Baseline (after 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 91 (9) | 88 (15)

10. Primary Outcome: Quality of Distance Vision
Description: as for outcome 9
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 87 (16) | 90 (12)

11. Primary Outcome: Quality of Near Vision
Description: Patient subjective scoring for quality of near vision using 0-100 continuous scale: 0=extremely poor vision all of the time. 100=excellent vision all of the time
Time Frame: Baseline (After 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 94 (8) | 91 (11)

12. Primary Outcome: Quality of Near Vision
Description: as for outcome 11
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 90 (12) | 90 (12)

13. Primary Outcome: Quality of Vision With Digital Device Use
Description: Subjective scoring of Quality of Vision with digital device use assessed using 0-100 continuous scale: (0=extremely poor vision all of the time. 100=excellent vision all of the time)
Time Frame: Baseline (After 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 96 (8) | 94 (7)

14. Primary Outcome: Quality of Vision With Digital Device Use
Description: as for outcome 13
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 91 (13) | 90 (12)

15. Primary Outcome: Quality of Intermediate Vision
Description: Subjective scoring of Quality of Intermediate Vision assessed using 0-100 continuous scale: (0=extremely poor vision all of the time. 100=excellent vision all of the time)
Time Frame: Baseline (After 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 97 (6) | 93 (9)

16. Primary Outcome: Quality of Intermediate Vision
Description: as for outcome 15
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 92 (11) | 92 (10)

17. Primary Outcome: Overall Vision Quality
Description: Subjective scoring of overall vision quality assessed using 0-100 continuous scale: (0=extremely poor vision all of the time. 100=excellent vision all of the time)
Time Frame: Baseline (After 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 95 (6) | 89 (13)

18. Primary Outcome: Overall Vision Quality
Description: as for outcome 17
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 88 (15) | 89 (12)

19. Secondary Outcome: Biomicroscopy Findings - Bulbar Hyperemia
Description: Bulbar hyperemia assessment using 5 categories: (0=None, 1= Slight injection to conjunctival vessels, 2= Mild injection, 3= Moderate injection, 4= Severe injection) in (0.25 steps)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 1.24 (0.67) | 1.37 (0.82)

20. Secondary Outcome: Biomicroscopy Findings- Limbal Hyperemia
Description: Investigator assessment using 5 categories: (0=None, 1= Slight injection to conjunctival vessels, 2= Mild injection, 3= Moderate injection, 4= Severe injection) in (0.25 steps)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 0.98 (0.69) | 1.21 (0.89)

21. Secondary Outcome: Biomicroscopy Findings - Corneal Staining Extent
Description: Investigator Assessment on Biomicroscopy Findings - Corneal Staining Extent on a scale of 0-4 : 0=No staining, 1=1-15% of area, 2=16-30% of area, 3=31-45% of area, 4= >45% of area
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale
  Central | 0.05 (0.21) | 0.10 (0.34)
  Nasal | 0.14 (0.34) | 0.16 (0.39)
  Temporal | 0.07 (0.26) | 0.03 (0.20)
  Superior | 0.13 (0.37) | 0.19 (0.40)
  Inferior | 0.34 (0.58) | 0.51 (0.74)

22. Secondary Outcome: Ghosting - Distance Vision
Description: Patient subjective scoring using 0-100 continuous scale:0=Intolerable;100=Not noticable
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 93 (12) | 93 (12)

23. Secondary Outcome: Ghosting - Near Vision
Description: Patient subjective scoring using 0-100 continuous scale:0=Intolerable;100=Not noticable
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 93 (10) | 93 (10)

24. Secondary Outcome: Overall Comfort
Description: Patient subjective scoring using 0-100 continuous scale, 0= cannot be worn, 100= cannot be felt ever.
Time Frame: Baseline (After 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 91 (8) | 89 (12)

25. Secondary Outcome: Overall Comfort
Description: Patient subjective scoring for overall comfort using 0-100 continuous scale, 0= cannot be worn, 100= cannot be felt ever.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 78 (23) | 79 (19)

26. Secondary Outcome: Overall Dryness
Description: Patient subjective scoring for overall dryness using 0-100 continuous scale, 0=cannot be worn, 100=no dryness experienced at any time.
Time Frame: Baseline (after 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 92 (12) | 92 (12)

27. Secondary Outcome: Overall Dryness
Description: as for outcome 26
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
Number analyzed (Participants) | 44 | 44
units on a scale | 76 (23) | 77 (21)

28. Secondary Outcome: Lens Preference - Overall Vision Preference
Description: Subjective rating of lens preference for overall vision preference (Phenacite, comfilcon A, No preference)
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 44
Participants
  Phenacite | 14
  comfilcon A | 25
  No Preference | 5

29. Secondary Outcome: Subjective Ratings of Change in Frequency of Tiredness
Description: Subjective rating of change in eye fatigue frequency of tiredness assessed using Eye fatigue Experience Questionnaire (EFEG)
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Groups:
- Phenacite: Subjects were randomized to wear phenacite study lens for one week.
  Phenacite: contact lens
- Comfilcon A: Subjects were randomized to wear comfilcon A contact lens for one week.
  comfilcon A : contact lens
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Much Better | 11 | 18
  Better | 50 | 39
  No Difference | 36 | 39
  Worse | 0 | 4
  Much Worse | 4 | 0

30. Secondary Outcome: Subjective Ratings of Change in Severity of Tiredness
Description: Subjective rating of change in eye fatigue severity of tiredness assessed using Eye fatigue Experience Questionnaire (EFEG)
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Much Better | 17 | 17
  Better | 48 | 39
  No Difference | 26 | 35
  Worse | 4 | 9
  Much Worse | 4 | 0

31. Secondary Outcome: Subjective Ratings of Change in Bothersome Rating for Tiredness
Description: Subjective rating of change in eye fatigue bothersome rating for tiredness assessed using Eye fatigue Experience Questionnaire (EFEG)
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Much Better | 20 | 10
  Better | 45 | 45
  No Difference | 35 | 40
  Worse | 0 | 5
  Much Worse | 0 | 0

32. Secondary Outcome: Subjective Ratings of Change in Frequency of Dryness
Description: Subjective rating of change in eye fatigue frequency of dryness assessed using Eye fatigue Experience Questionnaire (EFEG)
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Much Better | 15 | 20
  Better | 35 | 15
  No Difference | 25 | 35
  Worse | 15 | 25
  Much Worse | 10 | 5

33. Secondary Outcome: Subjective Ratings of Change in Severity of Dryness
Description: Subjective rating of change in eye fatigue severity of dryness assessed using Eye fatigue Experience Questionnaire (EFEG)
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Much Better | 9 | 5
  Better | 41 | 41
  No Difference | 32 | 27
  Worse | 9 | 23
  Much Worse | 9 | 5

34. Secondary Outcome: Subjective Ratings of Change in Bothersome Rating of Dryness
Description: Subjective rating of change in eye fatigue bothersome rating for dryness assessed using Eye fatigue Experience Questionnaire (EFEG)
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Much Better | 15 | 10
  Better | 40 | 40
  No Difference | 25 | 25
  Worse | 15 | 20
  Much Worse | 5 | 5

35. Secondary Outcome: Subjective Questionnaire Response - Eye Strain
Description: Subjective questionnaire response for " My eyes don't feel strained while wearing these lenses" - Agree, Disagree
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Agree | 75 | 75
  Disagree | 25 | 25

36. Secondary Outcome: Subjective Questionnaire Response - Eye Feel Good
Description: Subjective questionnaire response for " These lenses make my eyes feel good" - Agree, Disagree
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Agree | 86 | 71
  Disagree | 14 | 29

37. Secondary Outcome: Subjective Questionnaire Response - Eye Feel Relaxed
Description: Subjective questionnaire response for " These lenses make my eyes feel relaxed" - Agree, Disagree
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Agree | 79 | 79
  Disagree | 21 | 21

38. Secondary Outcome: Subjective Questionnaire Response - Vision
Description: Subjective questionnaire response for " These lenses help my vision" - Agree, Disagree
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Agree | 96 | 96
  Disagree | 4 | 4

39. Secondary Outcome: Subjective Questionnaire Response - Eye Tired
Description: Subjective questionnaire response for " These lenses make my eyes feel less tired" - Agree, Disagree
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Arm/Group | Phenacite | Comfilcon A
Number analyzed (Participants) | 44 | 44
percentage of participants
  Agree | 82 | 75
  Disagree | 18 | 25

ADVERSE EVENTS:
Time Frame: From dispense up to one week on each study lenses, a total of two weeks
Groups:
- Phenacite Test Lens: Participants were randomized to wear Phenacite test lens for one week.
  Phenacite: contact lens
- Comfilcon A Control Lens: Participants were randomized to wear comfilcon A control lens for one week.
  comfilcon A: contact lens
Arm/Group | Phenacite Test Lens | Comfilcon A Control Lens
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No